CLINICAL TRIAL: NCT00276341
Title: Efficacy of EGb 761® 120mg Twice a Day Versus Placebo on Cognitive Impairment in Patients With Multiple Sclerosis. A Randomised, Double-blind, Multicentre, Parallel Groups Placebo Controlled Phase III Study.
Brief Title: Study on the Effectiveness of EGb 761® vs Placebo Used for Cognitive Impairment in Patients With Multiple Sclerosis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ipsen (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2-39-00240-126
Record Dates: First submitted 2006-01-12; First posted 2006-01-13 (Estimated); Last update posted 2024-03-07 (Actual); Status verified 2024-03

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting
Keywords: cognitive impairment
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Cognitive Dysfunction | interventions — Ginkgo biloba extract

INTERVENTIONS:
Drug: EGb 761® (Tanakan®)

SUMMARY:
The purpose of this study is to determine whether the use of EGb 761 by patients with Relapsing-Remitting Multiple Sclerosis is effective in improving cognition, when compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Patient with Multiple Sclerosis Relapsing-Remitting form
* Patient with cognitive impairment (as spontaneous complaint by either patient or family)
* Patient treated with interferon and maintaining same dosage for previous 6 months
* Patient without major disability (Kurtzke Extended Disability Status Scale ≤6)

Exclusion Criteria:

* Clinical Multiple Sclerosis relapse within 3 months prior to participation
* Major psychiatric disease according to Diagnostic and Statistical Manual of Mental Disorders, 4th Ed.
* Other concomitant disorders possibly jeopardizing the cognitive status evaluation or the follow up of the patient (severe impairment of visual or motor function which may prevent participation in neuropsychological testing)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2003-08-26 (Actual); Study Completion 2005-12-08 (Actual)

PRIMARY OUTCOMES:
Evolution of Paced Auditory Serial Addition Test 3 and 2 seconds between baseline and week 24

SECONDARY OUTCOMES:
Evolution of the following tests between baseline and week 24:
Multiple Sclerosis Functional Composite Test
Selective Reminding Test
10/36 Visual-Spatial Recall Test
Symbol Digit Modalities Test
Trail Making Test A and B
Verbal Fluency Test
Empan Test
Evolution of the following scales between baseline and week 24:
Cognitive Deficit Interview based screen
Anxiety Brief Scale
Beck Depression Inventory Scale
Modified Fatigue Impact Scale
Evolution of Quality of Life
Evolution of the following between baseline, week 12, and week 24: Kurtzke Extended Disability Status Scale, and Clinician Interview Based Impression of Change

CONTACTS AND LOCATIONS:
Overall Officials: Ipsen Medical Director, Study Director — Ipsen
Locations (30):
- France (30):
  - Centre Hospitalier du Pays d'Aix, Aix-en-Provence
  - Hôpital Nord - CHU d'Amiens, Amiens
  - Hôpital J. Minjoz, Besançon
  - CHU de Bordeaux, Bordeaux
  - Groupe Hospitalier Pellegrin, Bordeaux
  - Hôpital de la cavale Blanche, Brest
  - Hôpital Neurologique, Bron
  - Hopital Nord, Cébazat
  - CHU Hôpital Gabriel Montpied, Clermont-Ferrand
  - Hôpital Civil de Colmar, Colmar
  - Hôpital Henri Mondor, Créteil
  - 14 bis Rue du Chapeau Rouge, Dijon
  - CHG Dijon, Dijon
  - Centre Hospitalier, Gonesse
  - Hôpital Universitaire Dupuytren, Limoges
  - Centre Hospitalier François, Mantes-la-Jolie
  - Hôpital Saint Joseph, Marseille
  - Hôpital Gui de Chauliac, Montpellier
  - Hôpital Central, Nancy
  - Hôpital Guillaume et Réne, Nantes
  - Hôpital Pasteur, Nice
  - Hôpital Léopold Bellan, Paris
  - Hôpital Saint Joseph, Paris
  - Centre Hospitalier René Dubos, Pontoise
  - Hôpital Laënnec, Quimper
  - CHU de Reims - Hôpital Maison Blanche, Reims
  - CHU Hôpital de Pontchaillou, Rennes
  - Hôpital Charles Nicolle, Rouen
  - Cabinet Médical, Rouen
  - Hôpital Delafontaine, Saint-Denis